CLINICAL TRIAL: NCT04072068
Title: A Phase IV Study on Impact of Edoxaban Treatment in Italian Cancer Patients With Venous Thromboembolism (EDOI Cancer Study) During Antineoplastic Therapy
Brief Title: Study on Impact of Edoxaban Treatment in Cancer Patients With Venous Thromboembolism During Antineoplastic Therapy
Acronym: EDOI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-05-2018
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Thromboembolism; Cancer
MeSH Terms: conditions — Thromboembolism; Neoplasms | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Edoxaban (Experimental): edoxaban 60 mg daily
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Every patient will receive every day edoxaban orally once a day. Edoxaban therapy will start after at least 5 days of lead-in with low-molecular-weight heparin, as per clinical practice. Edoxaban will be administered at dosage of 60 mg/day. In case of patients with body weight ≤60kg or with renal failure (creatinine clearance between 15 and 50 ml/min) or that are treated with P-gp inhibitors (cyclosporine, dronedarone, erythomycin, ketoconazole), dosage will be 30 mg/day. Patients will be treated for 6 up to 12 months with edoxaban, as per medical decision.

SUMMARY:
This is a multicentric, phase IV study. In this study patients that are receiving an antineoplastic treatment and that have been diagnosed with venous thromboembolism will receive edoxaban as per clinical practice. Edoxaban will be administered according to summary of product characteristics. Patients will receive 6 to 12 months of treatment with edoxaban administered orally. The thromboembolic event will be monitored as per local clinical practice. In this study patients will be evaluated at baseline, at the beginning of therapy with edoxaban, after 1 month (+/- 7 days), after 3, 6 and 12 months (+/- 3 weeks). During these visits, patients will be provided of a diary in which they should report drug intake and interruptions and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects presenting with VTE (venous thromboembolism) associated with cancer (other than basal-cell or squamous-cell carcinoma of the skin). Cancer diagnosis should be done within two years prior to VTE.
* Patient must be receiving systemic antineoplastic therapy (such as chemotherapy, target therapy, immunotherapy, hormonotherapy) and remain candidate to receive at least other 3 months of anti neoplastic therapy.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients;
* Clinically significant active bleeding;
* Hepatic disease associated with coagulopathy and clinically relevant bleeding risk;
* Lesion or condition, if considered to be a significant risk for major bleeding. This may include current or recent gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial haemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities;
* Uncontrolled severe hypertension;
* Concomitant treatment with any other anticoagulants
* Pregnancy and breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of edoxaban related adverse events on antineoplastic therapy | 24 months
  Percentage of antineoplastic therapy delays/interruption due to ADR related to edoxaban (bleeding, hepatobiliary toxicity, renal toxicity, anemia, hypersensitivity reactions).
Quality of life questionnaire | 24 months
  Quality of life will be evaluated using validate quality of life questionnaires.

SECONDARY OUTCOMES:
Evaluate the compliance to Edoxaban treatment | 24 months
  For every patient the number of edoxaban tables used will be assessed and compared with the prescribed dose.
Evaluate the safety of edoxaban treatment | 24 months
  The adverse event severity grading scale for the National Cancer Institute Common Terminology for Adverse Events, Version 4.0 (NCI CTCAE v4.0) will be used for assessing adverse event severity.

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Pinto, MD, Principal Investigator — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (18):
- Italy (18):
  - Presidio Ospedaliero SS. Antonio e Biagio, Alessandria
  - Istituto Tumori di Bari, Bari
  - Azienda Ospedalier Spedali Civili di Brescia, Brescia
  - Ospedale S.Giacomo, Castelfranco Veneto
  - ARNAS Garibaldi, Catania
  - Istituti Ospitalieri di Cremona, Cremona
  - Ospedale di Faenza, Faenza
  - Ospedale Civile di Guastalla, Guastalla
  - Ospedale Mater Salutis, Legnago
  - Istituto Nazionale dei Tumori di Milano, Milan
  - Ospedali Monaldi Cotugno, Napoli
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - AUSL/IRCCS di Reggio Emilia, Reggio Emilia
  - Ospedale degli Infermi, Rimini
  - ASST Valleolona, PO Saronno, Saronno
  - Ospedale Mauriziano, Torino
  - Ospedale Molinette, Torino

IPD SHARING:
Plan to Share IPD: No